CLINICAL TRIAL: NCT05788432
Title: Sequent Please Neo Extended Post-Market Clinical Follow-up Study
Brief Title: Sequent Extended Study
Acronym: rEpic06
Status: Recruiting | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: rEpic06- SEQUENT EXTENDED
Record Dates: First submitted 2023-03-13; First posted 2023-03-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease
Keywords: MDR (Medical Device Regulations); PMCF (Post-Market Clinical Follow-up); Paclitaxel eluting coronary balloon dilatation catheter
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Disease (CAD)
  Interventions: Device: Sequent Please Neo

INTERVENTIONS:
Device: Sequent Please Neo — Patients in whom treatment with (Sequent Please Neo) has been attempted

SUMMARY:
Multicenter, prospective, non-randomized, post-market clinical follow-up (PMCF) study to confirm and support the clinical safety and performance of Sequent Please Neo to meet EU Medical Device regulation (MDR) requirements in all the consecutive patients treated with Sequent Please Neo.

DETAILED DESCRIPTION:
The objective of this multicenter, prospective, non-randomized, postmarket clinical follow-up(PMCF) study is to confirm and support the clinical safety and performance of the Sequent Please Neo in a NON-SELECTED, Real Word population under daily clinical practice when used as intended by the manufacturer to meet EU Medical Device Regulation requirements for post-market clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with Sequent please neo according to routine hospital practice and following instruction for use.
* Informed Consent Signed.

Exclusion Criteria:

* Patient life expectancy less than 12 months.
* Contraindication for antiplatelet therapy.
* Not meet inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Sequent Please Neo according to routine hospital practice and following instructions for use.
Sampling Method: Non-Probability Sample
Enrollment: 2028 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety & Effectiveness. Freedom from MACE (Major Adverse Cardiac Events) | 12 months
  Composite endpoint of death, myocardial infarction (MI) and a new Target Lesion Revascularization (TLR)

SECONDARY OUTCOMES:
Freedom from MACE in the subgroup of Lesions In-stent Restenosis | 12 months
  Freedom from MACE in the subgroup of Lesions In-stent Restenosis
Freedom from MACE in the subgroup of Native vessel lesions | 12 months
  Freedom from MACE in the subgroup of Native vessel lesions
Freedom from MACE in the subgroup of Lesions in Bifurcation Side Branches | 12 months
  Freedom from MACE in the subgroup of Lesions in Bifurcation Side Branches
Procedural success | Immediately after PCI (Percutaneous Coronary Intervention)
  Procedural success ( Residual stenosis <30% and absence of dissection and TIMI ( Thrombolysis in Myocardial Infarction) flow 3 after procedure)

CONTACTS AND LOCATIONS:
Locations (26):
- Spain (26):
  - Hospital Universitario de Araba, Alava
  - Hospital General Universitario de Alicante Dr.Balmis, Alicante
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital de La Santa Creu Y Sant Pau, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Puerta Del Mar, Cadiz
  - Hospital General Universitari de Castelló, Castelló
  - Hospital Universitario San Pedro de Alcantara, Cáceres
  - Hospital Universitario de Ciudad Real, Ciudad Real
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitario de Cabueñes, Gijón
  - Hospital Universitari Dr. Josep Trueta, Girona
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitario de Jaen, Jaén
  - Hospital Universitario de Leon, León
  - Hospital Universitario Lucus Agusti, Lugo
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen de La Victoria, Málaga
  - Hospital de Mérida, Mérida
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital General Universitario de Toledo, Toledo

REFERENCES:
- [Background] Rissanen TT, Uskela S, Eranen J, Mantyla P, Olli A, Romppanen H, Siljander A, Pietila M, Minkkinen MJ, Tervo J, Karkkainen JM; DEBUT trial investigators. Drug-coated balloon for treatment of de-novo coronary artery lesions in patients with high bleeding risk (DEBUT): a single-blind, randomised, non-inferiority trial. Lancet. 2019 Jul 20;394(10194):230-239. doi: 10.1016/S0140-6736(19)31126-2. Epub 2019 Jun 13. PMID 31204115
- [Background] Jeger RV, Farah A, Ohlow MA, Mangner N, Mobius-Winkler S, Leibundgut G, Weilenmann D, Wohrle J, Richter S, Schreiber M, Mahfoud F, Linke A, Stephan FP, Mueller C, Rickenbacher P, Coslovsky M, Gilgen N, Osswald S, Kaiser C, Scheller B; BASKET-SMALL 2 Investigators. Drug-coated balloons for small coronary artery disease (BASKET-SMALL 2): an open-label randomised non-inferiority trial. Lancet. 2018 Sep 8;392(10150):849-856. doi: 10.1016/S0140-6736(18)31719-7. Epub 2018 Aug 28. PMID 30170854
- [Background] Alfonso F, Perez-Vizcayno MJ, Cardenas A, Garcia del Blanco B, Garcia-Touchard A, Lopez-Minguez JR, Benedicto A, Masotti M, Zueco J, Iniguez A, Velazquez M, Moreno R, Mainar V, Dominguez A, Pomar F, Melgares R, Rivero F, Jimenez-Quevedo P, Gonzalo N, Fernandez C, Macaya C; RIBS IV Study Investigators (under auspices of Interventional Cardiology Working Group of Spanish Society of Cardiology). A Prospective Randomized Trial of Drug-Eluting Balloons Versus Everolimus-Eluting Stents in Patients With In-Stent Restenosis of Drug-Eluting Stents: The RIBS IV Randomized Clinical Trial. J Am Coll Cardiol. 2015 Jul 7;66(1):23-33. doi: 10.1016/j.jacc.2015.04.063. PMID 26139054
- [Background] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. N Engl J Med. 2006 Nov 16;355(20):2113-24. doi: 10.1056/NEJMoa061254. Epub 2006 Nov 13. PMID 17101615
- [Background] Unverdorben M, Kleber FX, Heuer H, Figulla HR, Vallbracht C, Leschke M, Cremers B, Hardt S, Buerke M, Ackermann H, Boxberger M, Degenhardt R, Scheller B. Treatment of small coronary arteries with a paclitaxel-coated balloon catheter. Clin Res Cardiol. 2010 Mar;99(3):165-74. doi: 10.1007/s00392-009-0101-6. Epub 2010 Jan 6. PMID 20052480